CLINICAL TRIAL: NCT00094640
Title: Pharmacokinetic Characterization of Intramuscular Olanzapine Depot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 6106; F1D-EW-LOBS
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: Intramuscular Olanzapine Depot

SUMMARY:
The goals of this study are to:

Determine the blood levels of intramuscular (IM) olanzapine depot in patients at different points in time after an injection, and compare these levels to the amount of olanzapine in the blood of patients after treated by oral administration with Zyprexa (olanzapine) tablets or by intramuscular administration with Zyprexa IntraMuscular (olanzapine for injection).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have schizophrenia or schizoaffective disorders.
* Each patient must have a level of understanding sufficient to complete all tests and examinations required by the protocol, and to provide informed consent.
* Patient must not have participated in a clinical trial of another investigational drug, including olanzapine, within 1 month (30 days) prior to study entry.
* Female patients must not be pregnant or breast-feeding.
* Patients must not be experiencing acute, serious, or unstable medical conditions other than schizophrenia or schizoaffective disorder.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Adelaide, South Australia, Australia
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kortenberg, Belgium
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Rio de Janeiro, Rio de Janeiro, Brazil
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Zagreb, Croatia
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Prague, Czechia
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mexico City, Tlalpan, Mexico
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bratislava, Slovakia
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Barcelona, Spain

REFERENCES:
- [Derived] Atkins S, Detke HC, McDonnell DP, Case MG, Wang S. A pooled analysis of injection site-related adverse events in patients with schizophrenia treated with olanzapine long-acting injection. BMC Psychiatry. 2014 Jan 14;14:7. doi: 10.1186/1471-244X-14-7. PMID 24423017
- [Derived] McDonnell DP, Detke HC, Bergstrom RF, Kothare P, Johnson J, Stickelmeyer M, Sanchez-Felix MV, Sorsaburu S, Mitchell MI. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, II: investigations of mechanism. BMC Psychiatry. 2010 Jun 10;10:45. doi: 10.1186/1471-244X-10-45. PMID 20537130
- [Derived] Detke HC, McDonnell DP, Brunner E, Zhao F, Sorsaburu S, Stefaniak VJ, Corya SA. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, I: analysis of cases. BMC Psychiatry. 2010 Jun 10;10:43. doi: 10.1186/1471-244X-10-43. PMID 20537128